CLINICAL TRIAL: NCT02742064
Title: Quantified Mobile Sensing for Improving Diagnosis and Measuring Disease Progression
Status: Completed | Type: Observational
Sponsor: Cogito Health Inc (Industry)
Collaborators: Massachusetts General Hospital (Other); Partners HealthCare (Other)
Responsible Party: Sponsor
Other Study IDs: 1R44MH107065-01 (NIH)
Record Dates: First submitted 2016-04-11; First posted 2016-04-18 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Depression; Bipolar Disorder
MeSH Terms: conditions — Depression; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MDD-Single Episode: 1. Subjects who have experienced 1 episode of major depressive disorder (MDD) in their lifetime.
  Interventions: Other: Cogito Companion Mobile Phone Application
- MDD-Recurrent: 1. Subjects who have experienced 2 or more episodes of depressive disorder (MDD) in their lifetime.
  Interventions: Other: Cogito Companion Mobile Phone Application
- Bipolar Disorder: 1. Subjects who have been diagnosed with bipolar disorder in their lifetime.
  Interventions: Other: Cogito Companion Mobile Phone Application

INTERVENTIONS:
Other: Cogito Companion Mobile Phone Application
  Other Names: Cogito Mobile Sensing Platform

SUMMARY:
The purpose of this study is to determine if a mobile sensing platform can passively and objectively detect the presence of clinically significant mood disorder symptomatology and symptom progression over time. Meeting this goal will allow for improved risk categorization, prediction of relapse, and measurement of disease progression in a lifetime prevalence population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Have a smartphone and cell service plan, including voice and data, that meets the device requirements of the Mobile Sensing Platform.
* Enrolled in the MoodNetwork

Exclusion Criteria:

* Report positively on the QIDS-SR suicide item during study intake
* Total score greater than 15 on the QIDS-SR during the screening process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the MoodNetwork, an online network of individuals with mood disorders, which is hosted by MGH. A subset of participants with mood disorders enrolled in MoodNetwork will download Cogito's mobile sensing platform on their mobile phones.
Sampling Method: Non-Probability Sample
Enrollment: 899 (Actual)
Dates: Start 2015-02; Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Severity of MDD symptoms as assessed by QIDS SR | 6 months
Severity of Mania symptoms as assessed by ASRM | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No